CLINICAL TRIAL: NCT00597883
Title: Neurologic and Neuropsychometric Outcome in Patients Undergoing Carotid Endarterectomy
Brief Title: Neuropsychometric Outcome After Carotid Endarterectomy
Acronym: CEA
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAA4811
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Results first posted 2024-12-03 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Carotid Artery Stenosis; Carotid Artery Disease; Transient Ischemic Attack; Stroke
Keywords: carotid endarterectomy; Neuropsychological tests; Stroke; Transient ischemia
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases; Ischemic Attack, Transient; Stroke | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum plasma DNA (via buccal samples will be obtained using a buccal cell collection swab)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients having CEA: Patients undergoing carotid endarterectomy (CEA) for treatment of carotid artery stenosis will receive neurological and neuropsychological evaluations
  Interventions: Procedure: Carotid endarterectomy; Other: Neurological and neuropsychological evaluations

INTERVENTIONS:
Procedure: Carotid endarterectomy — (non-experimental) carotid endarterectomy (CEA) for treatment of carotid artery stenosis
Other: Neurological and neuropsychological evaluations — Clinical examinations consisting of a neurological and neuropsychological evaluation

SUMMARY:
The purpose of this study is to determine how well patients undergoing carotid endarterectomy will perform on a battery of tests to assess brain function before and after surgery as compared to a control group of patients undergoing spine surgery. This study will serve to: (a) determine incidence of neurologic/neuropsychometric change in patients undergoing carotid artery surgery, and (b) to ascertain the time it takes for these changes to resolve.

DETAILED DESCRIPTION:
Cerebral injury will be determined in four ways. First, all patients will be evaluated using a battery of neuropsychometric tests before and after surgery. Patients admitted to the Irving Clinical Research Center (CRC) will have their tests one day before, one day after surgery and at 1 month. Those coming into the hospital on the day of surgery, "Same Day", will be evaluated on the day of surgery, one day after and at the 1 month follow up. Preoperative neurological and neuropsychological evaluation will be performed. The neuropsychometric tests are not intended to be diagnostic of specific neuropsychiatric disorders, but rather are designed to demonstrate general neuropsychological pathology. These tests can be divided into four types: (1) an evaluation of language, (2) an evaluation of speed of mental processing, (3) an evaluation of ability to learn using a list of words, and (4) an evaluation of visual perception requiring a patient to copy a complex figure. Before the battery is administered we will assess each patient's level of pain while sitting and standing using a 10 point Visual Analog Scale and then gauge their mood with a series called the Wong/Baker Faces Rating scale.

We will be measuring Quality of Life (QOL) in all enrolled patients. This will be done using two well-known examinations (Telephone Interview for Cognitive Status (TICS) and Centers for Disease Control and Prevention Health-Related Quality of Life 14 Item Measure (CDC HRQOL14)) and a series of questions investigating how well patients are able to perform activities of daily living (ADLs) and instrumental activities of daily living (IADLs). These tests will be given at two time points, once before the surgery and then one month after surgery. We will look for changes in quality of life that may correlate with neuropsychometric test performance.

Peripheral serum samples will be drawn before induction, before cross-clamping the carotid artery, 15 minutes after cross-clamping the carotid artery and 24 hours after surgery. These samples will be analyzed for four different sets of markers of cerebral injury, one gene and two markers of systemic inflammation. Serum levels of neuron specific enolase (NSE) and protein S100B, a neuronal enzyme and glial cell component respectively, markers of cell injury will demonstrate cerebral injury

Patients will undergo intraoperative TCD (Transcranial Doppler) The TCD examination will assess the brain's ability to increase cerebral blood flow in response to a pharmacological challenge (CO2 inhalation). TCD measures the degree of cerebral vasodilation, identified as an increase in flow velocity on TCD. This "cerebrovascular reserve" we hypothesize will be able to predict performance on postoperative neuropsychometric tests

ELIGIBILITY:
Inclusion Criteria:

* ability to speak English
* undergoing carotid endarterectomy procedure
* undergoing lumbar laminectomy procedure

Exclusion Criteria:

* history of permanent neurological impairment
* Axis I psychiatric diagnosis or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Columbia University/NY Presbyterian Hospital
Sampling Method: Non-Probability Sample
Enrollment: 817 (Actual)
Dates: Start 2003-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Heyer, M.D., Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University, Department of Anesthesiology, New York, New York, United States

REFERENCES:
- [Background] Parsson HN, Lord RS, Scott K, Zemack G. Maintaining carotid flow by shunting during carotid endarterectomy diminishes the inflammatory response mediating ischaemic brain injury. Eur J Vasc Endovasc Surg. 2000 Feb;19(2):124-30. doi: 10.1053/ejvs.1999.0954. PMID 10727360
- [Background] Jaranyi Z, Szekely M, Bobek I, Galfy I, Geller L, Selmeci L. Impairment of blood-brain barrier integrity during carotid surgery as assessed by serum S-100B protein concentrations. Clin Chem Lab Med. 2003 Oct;41(10):1320-2. doi: 10.1515/CCLM.2003.201. PMID 14580159
- [Background] Hetzel A, Braune S, Guschlbauer B, Dohms K. CO2 reactivity testing without blood pressure monitoring? Stroke. 1999 Feb;30(2):398-401. doi: 10.1161/01.str.30.2.398. PMID 9933278
- [Background] Valdueza JM, Draganski B, Hoffmann O, Dirnagl U, Einhaupl KM. Analysis of CO2 vasomotor reactivity and vessel diameter changes by simultaneous venous and arterial Doppler recordings. Stroke. 1999 Jan;30(1):81-6. doi: 10.1161/01.str.30.1.81. PMID 9880393
- [Result] Heyer EJ, Adams DC, Solomon RA, Todd GJ, Quest DO, McMahon DJ, Steneck SD, Choudhri TF, Connolly ES. Neuropsychometric changes in patients after carotid endarterectomy. Stroke. 1998 Jun;29(6):1110-5. doi: 10.1161/01.str.29.6.1110. PMID 9626280
- [Result] Heyer EJ, Mergeche JL, Bruce SS, Connolly ES. Inflammation and cognitive dysfunction in type 2 diabetic carotid endarterectomy patients. Diabetes Care. 2013 Oct;36(10):3283-6. doi: 10.2337/dc12-2507. Epub 2013 Jun 4. PMID 23735728
- [Result] Heyer EJ, Mergeche JL, Ward JT, Malone HR, Kellner C, Bruce SS, Connolly ES. Phosphodiesterase 4D single-nucleotide polymorphism 83 and cognitive dysfunction in carotid endarterectomy patients. Neurosurgery. 2013 Nov;73(5):791-6; discussion 796. doi: 10.1227/NEU.0000000000000085. PMID 23863764
- [Result] Heyer EJ, Mergeche JL, Bruce SS, Ward JT, Stern Y, Anastasian ZH, Quest DO, Solomon RA, Todd GJ, Benvenisty AI, McKinsey JF, Nowygrod R, Morrissey NJ, Connolly ES. Statins reduce neurologic injury in asymptomatic carotid endarterectomy patients. Stroke. 2013 Apr;44(4):1150-2. doi: 10.1161/STROKEAHA.111.000362. Epub 2013 Feb 12. PMID 23404722
- [Result] Heyer EJ, Kellner CP, Malone HR, Bruce SS, Mergeche JL, Ward JT, Connolly ES Jr. Complement polymorphisms and cognitive dysfunction after carotid endarterectomy. J Neurosurg. 2013 Sep;119(3):648-54. doi: 10.3171/2013.4.JNS1368. Epub 2013 May 10. PMID 23662819
- [Derived] Heyer EJ, Mergeche JL, Wang S, Gaudet JG, Connolly ES. Impact of Cognitive Dysfunction on Survival in Patients With and Without Statin Use Following Carotid Endarterectomy. Neurosurgery. 2015 Dec;77(6):880-7. doi: 10.1227/NEU.0000000000000904. PMID 26308635
- [Derived] Sussman ES, Kellner CP, Mergeche JL, Bruce SS, McDowell MM, Heyer EJ, Connolly ES. Radiographic absence of the posterior communicating arteries and the prediction of cognitive dysfunction after carotid endarterectomy. J Neurosurg. 2014 Sep;121(3):593-8. doi: 10.3171/2014.5.JNS131736. Epub 2014 Jul 4. PMID 24995780
- [Derived] Halazun HJ, Mergeche JL, Mallon KA, Connolly ES, Heyer EJ. Neutrophil-lymphocyte ratio as a predictor of cognitive dysfunction in carotid endarterectomy patients. J Vasc Surg. 2014 Mar;59(3):768-73. doi: 10.1016/j.jvs.2013.08.095. PMID 24571940
- [Derived] Heyer EJ, Mergeche JL, Connolly ES Jr. Middle cerebral artery pulsatility index and cognitive improvement after carotid endarterectomy for symptomatic stenosis. J Neurosurg. 2014 Jan;120(1):126-31. doi: 10.3171/2013.8.JNS13931. Epub 2013 Sep 6. PMID 24010976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients having CEA surgery were recruited independently of patients in the reference group, who were having "simple" spine surgery. Therefore, the 155 patients having "simple" spine surgery were not double counted.
Groups:
- CEA Patients: Consecutive patients were enrolled who were having elective carotid endarterectomy. Performance in these patients were based on testing before and after CEA at two time points: one and thirty days after surgery. The difference in performance on a battery of neuropsychometric tests was scored by comparing the mean and standard deviation in the change scores to a reference consisting of patients having "simple" spine surgery defined as microdiskectomy or one or two level laminectomies lasting less than four hours, not requiring blood transfusions and not needing to be admitted to the intensive care unit.
- Reference Group: Patients had "simple" spine surgery instead of Carotid endarterectomy
Period: Overall Study
Arm/Group | CEA Patients | Reference Group
Started | 662 (The total number of patients (CEA and Reference) was 817, 662 CEA and 155 reference.) | 155 (The reference group was not part of another study. They were recruited for this study only.)
Completed | 662 (Total number of patients tested were 662. About 900 patients approached.) | 155
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CEA Patients | Reference Group | Total
Number analyzed (Participants) | 662 | 155 | 817
Age, Customized [Mean (Full Range); unit: years] — The mean and full range of the total is verified.
  years
    Age | 72 [50 to 90] | 71 [70 to 72] | 72 [50 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 232 | 55 | 287
  Male | 430 | 100 | 530
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 0 | 42
  Not Hispanic or Latino | 18 | 0 | 18
  Unknown or Not Reported | 602 | 155 | 757
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 0 | 18
  White | 578 | 0 | 578
  More than one race | 10 | 0 | 10
  Unknown or Not Reported | 52 | 155 | 207
Region of Enrollment [Number; unit: participants]
  United States | 662 | 155 | 817

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Having a Significant Change in Neuropsychometric Performance After Carotid Endarterectomy
Description: Neuropsychometric performance change is measured in Z-scores by compared to a reference group of elderly patients > 60 years having "simple" spine surgery. The Z-scores were generated as follows. The mean and standard deviation (SD) of the change scores (neurocognitive performance after surgery minus neurocogntivie performance before surgery [baseline]) was calculated for the reference group of patients. The mean and SD from the reference group was used to generate Z-scores: The mean change score from the reference group of patients was subtracted from the change scores in for each CEA patient for each test and divided by the SD of the change scores of the reference group of patients.
Time Frame: Baseline to Day 1
Measure: Number; unit: percentage of participants
Groups:
- Reference Group: Patients had spine surgery
Arm/Group | CEA Patients | Reference Group
Number analyzed (Participants) | 662 | 155
percentage of participants | 22 | 4.5

ADVERSE EVENTS:
Time Frame: 11 years
Description: All patients were examined with a battery of neuropsychometric tests before and after having carotid endarterectomy surgery.
Arm/Group | Reference Group | CEA Patients
All-Cause Mortality (participants affected / at risk) | 0/155 | 0/662
Serious Adverse Events (participants affected / at risk) | 0/155 | 0/662
Other Adverse Events (participants affected / at risk) | 0/155 | 12/662
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reference Group (N=155) | CEA Patients (N=662)
Stroke (Vascular disorders) | 0 (0) | 12 (12) — Stroke, which occurred in 12 patients. Stroke was defined as a new neurologic finding.

LIMITATIONS AND CAVEATS:
Data for multiple time points (30 days) are inconclusive due to patient dropout. Data sets evolved between 1995-2012, and a master database linking subjects to publications was missing, obscuring sample derivation. Reported methods likely overstate neuropsychiatric testing completeness. Reasons for 'missingness' were multifactorial preventing assessment of impacts. Relevant journals were informed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No